CLINICAL TRIAL: NCT02370212
Title: Interval Training Plus Creatine Effects on Performance and Glucose Tolerance
Acronym: Cr + HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H15--00205
Record Dates: First submitted 2015-02-04; First posted 2015-02-24 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Creatine; interval training; effects on performance
MeSH Terms: interventions — Creatine; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Creatine (Experimental): Creatine will be ingested after interval training and at supper time on training days and in the morning and afternoon on non-training days (0.05 g/kg body mass of creatine with 0.05 g/kg flavoured dextrose per dose).
  Both experimental and placebo groups will perform the same high intensity interval training protocols (3x/week for 4 weeks).
  Interventions: Dietary Supplement: Creatine; Other: High intensity interval training
- Placebo (Placebo Comparator): The placebo will be ingested after interval training and at supper time on training days and in the morning and afternoon on non-training days (0.1 g/kg flavoured dextrose per dose, isocaloric to the creatine).
  Both experimental and placebo groups will perform the same high intensity interval training protocols (3x/week for 4 weeks).
  Interventions: Dietary Supplement: Placebo; Other: High intensity interval training

INTERVENTIONS:
Dietary Supplement: Creatine
  Arms: Creatine
Dietary Supplement: Placebo
  Arms: Placebo
Other: High intensity interval training

SUMMARY:
Recent evidence suggests that high -intensity interval training (HIIT) may be an effective strategy to improve cardiorespiratory fitness, exercise performance, and insulin sensitivity. In addition, creatine (Cr), a nitrogen- containing compound, is widely used to enhance high intensity exercise performance. A seminal study demonstrated that the muscle content of Cr and phosphocreatine (PCr) can be elevated by exogenous Cr. Oral intake of Cr increases the concentration in blood and muscle, and part of the increased muscle Cr is transformed to PCr (a process catalyzed by Cr kinase). Cr supplementation increases total Cr (TCr = Cr + PCr) by ~20%, with the PCr component accounting for 10% of the increase.

Combining HIIT and Cr is intriguing for two reasons; first, Cr supplementation improves performance through increasing PCr, PCr recovery, and muscle buffering which may facilitate higher training intensities and therefore greater training adaptations. Secondly, both Cr and HIIT have individually been shown to increase GLUT 4 and insulin sensitivity, suggesting that Cr supplementation may be an adjunct to HIIT for improving glucose control. To date, there have only been two studies investigating the performance effects of Cr combined with HIIT with preliminary positive results. No studies have examined the impact of combined Cr + HIIT on outcomes related to insulin sensitivity. Therefore, the purpose of this research is to examine the combined effects of Cr and HIIT on performance and insulin sensitivity as determined via an oral glucose tolerance test (OGTT) in young healthy adults.

DETAILED DESCRIPTION:
PURPOSE: To determine whether combining creatine with high intensity interval training (HIIT) results in better exercise performance and insulin sensitivity when compared to HIIT combined with placebo in healthy subjects.

HYPOTHESES: a) Creatine + HIIT will result in improved exercise performance compared to placebo; b) Creatine + HIIT will result in improved insulin sensitivity compared to placebo.

OBJECTIVES: To determine whether combining creatine with high intensity interval training (HIIT) results in better exercise performance and insulin sensitivity when compared to HIIT combined with placebo in healthy subjects.

RESEARCH METHOD: A double blind placebo randomized controlled trial (RCT) in which 24 healthy young volunteers will participate in HIIT three times a week, for four weeks. Participants will be will be stratified for sex and randomized to one of two interventions; 1) HIIT plus Cr, or 2) HIIT plus placebo.

STATISTICAL ANALYSES: A 2 (group) x 2 (time) way repeated measures ANOVA will be used to analyze all variables. Descriptive statistics (means, standard deviations [SD], and frequencies) will be calculated. Histograms will be used to identify any outliers and to test for normality. Data with skewed distributions will be log-transformed prior to statistical testing. Within group differences will be examined by paired t-test.

24 participants will be included in this RCT. Sample size calculations were computed using means and standard deviations from a previous Cr + HIIT study [11] which showed an significant increase in cycling critical power with Cr + HIIT (6.72 +/- 2.54 % increase) compared to Placebo + HIIT (3.82 +/- 2.30 %). With 80% power at an alpha of 0.05 indicated that 11 participants per group are needed. To preserve power and account for potential drop-out we will recruit 12 per group.

ELIGIBILITY:
Inclusion Criteria:

* Between 18--35 years of age
* Can read, comprehend, and speak English
* Free of diagnosed metabolic disease (e.g., prediabetes, diabetes)
* Willing and able to perform high-intensity exercise training
* Willing and able to consume creatine or placebo supplements over the study period

Exclusion Criteria:

* Diagnosed metabolic disorder such as diabetes, metabolic syndrome, prediabetes, hypothyroidism, cardiovascular disease or any other condition known to affect metabolism
* Currently engaged in high-intensity interval training >2 time per week
* Currently taking creatine or other supplements or having taken creatine in the last 12 weeks

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in exercise performance at 4 weeks | 4 weeks
  Assessed by a 50 kilojoule (kJ) time trial test

SECONDARY OUTCOMES:
Change from Baseline in cardiorespiratory fitness | 4 weeks
  Measured by a VO2peak test
Change from Baseline in body composition | 4 weeks
  Measured by a DXA scan
Change from Baseline in insulin sensitivity | 4 weeks
  Assessed using an oral glucose tolerance test (OGTT)